CLINICAL TRIAL: NCT05362175
Title: Comparison of the Efficacy Between Ultrasound Measurement of Cross Sectional Area of the Umbilical Cord and Hadlock's Formula in Prediction of Neonatal Birth Weight at Term Gestation:Cross Sectional Study
Brief Title: Cross Sectional Area of Umbilical Cord Versus Hadlock's Formula in Prediction of Neonatal Birth Weight
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mena shafeek Ibrahim ghaly, Mena Shafeek, Ain Shams University
Other Study IDs: Ain Shams University Hos
Record Dates: First submitted 2021-08-26; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Birth Weight; Fetal Body Weight
Keywords: Birth weight; Hadlock's formula; Cross sectional area of umbilical cord; Umbilical cord; Fetal biometry
MeSH Terms: conditions — Birth Weight; Fetal Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Cross sectional area of umbilical cord and Hadlock's formula: Ultrasound measurement of cross sectional area of umbilical cord within 1 cm from the umbilical cord insertion into the fetal abdomen And Fetal biometry using the standard Hadlock's formula
  Interventions: Device: Obstetric ultrasound

INTERVENTIONS:
Device: Obstetric ultrasound — ultrasound measurement of the cross sectional area of umbilical cord within 1 cm from the cord insertion in to fetal abdomen and the standard Hadlock's formula

SUMMARY:
Ultrasound measurement of cross sectional area of umbilical cord might offer advantage over Hadlock's formula for accurate estimation of actual birth weight at term gestation leading to prevention of large number of maternal and neonatal morbidity and mortality.

DETAILED DESCRIPTION:
Umbilical cord is a vital structure of maternal-fetal life that can be used to evaluate pregnancy outcomes. In the past, sonographic investigations of the umbilical cord were limited to identification of the number of vessels and Doppler evaluation of the blood flow. Various formulas have developed to calculate Estimated Fetal Weight (EFW) using fetal biometry. While it is being accurate to a degree, they are associated with error especially with extreme birth weight. In this study using the ultrasound to look for a relation between the umbilical cord cross sectional area and estimated birth weight, as it's easy to use and readily available, comparing the estimated birth weight obtained by this method with that of Hadlock's formula measures at term gestation. Trying to prove that the umbilical cord area formula might gave advocacy for future usage for birth weight prediction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with:

  * Age: 18-35 years.
  * Singleton living fetus.
  * Term gestation (37wks_ 41wks+6days). (Spong , 2013).
  * Admitted at labor room or prepared for caesarean section

Exclusion Criteria:

* o Intrauterine Dead fetus (IUFD).

  * Structurally malformed fetus or umbilical cord (single umbilical artery; SUA).
  * Multiple pregnancies.
  * Oligohydraminos (AFI < 5cm or DVP <2 cm) or polyhydraminos (AFI > 25 cm or DVP > 8 cm) (Morteza et al., 2018).
  * Uterine fibroid.
  * Abnormal Doppler flowmetry of umbilical artery.
  * Maternal diseases (Diabetes mellitus, Hypertensive disorders, renal diseases, Ischemic heart diseases), history of drug intake (Antihypertensive, antiepileptic, oral hypoglycemic drugs).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women at term gestation admitted at labor room or prepared for cesarean section
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Estimated fetal weight calculation by hadlock's formula and by umbilical cord cross sectional area ,then correlation with actual birth weight measured with in 1st hour of delivary | 1st hour of delivary
  correlation with actual birth weight measured

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No